CLINICAL TRIAL: NCT01254604
Title: A Phase III, Randomized, Active Comparator-Controlled, Four-Week, Double-Masked Clinical Trial to Compare the Efficacy and Safety of Preservative-Free MK-2452 (0.0015%) and Preservative-Free Timolol Maleate (0.5%) in Patients With Open-Angle Glaucoma or Ocular Hypertension in India
Brief Title: Preservative-Free Tafluprost (MK-2452) for the Treatment of Open-Angle Glaucoma or Ocular Hypertension (MK-2452-002)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2452-002
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Tafluprost; Glaucoma; Ocular Hypertension; Timolol; Eye Disorder; Preservative-Free; Prostaglandin Analogue
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tafluprost (Experimental): One drop of preservative-free vehicle (contains no active drug) per eye in the morning, and one drop of preservative-free tafluprost (0.0015%) per eye in the evening for four weeks. Morning dose with vehicle only allows blinding to match twice daily dosing of comparator arm.
  Interventions: Drug: Preservative-Free Tafluprost or vehicle
- Timolol (Active Comparator): One drop of preservative-free timolol maleate (0.05%) per eye twice daily (morning and evening) for four weeks.
  Interventions: Drug: Preservative-Free Timolol maleate

INTERVENTIONS:
Drug: Preservative-Free Tafluprost or vehicle — Preservative-free tafluprost (0.0015%) ophthalmic solution; Preservative-free vehicle ophthalmic solution (contains no active drug)
  Other Names: MK-2452
  Arms: Tafluprost
Drug: Preservative-Free Timolol maleate — Preservative-free timolol maleate (0.5%) ophthalmic solution
  Other Names: Preservative-Free Timoptic
  Arms: Timolol

SUMMARY:
This study will test the hypothesis that preservative-free tafluprost (MK-2452) is non-inferior to preservative-free timolol maleate with respect to the diurnal intraocular pressure (IOP) change from baseline after 4 weeks of therapy in participants with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participant has been diagnosed with primary open-angle glaucoma, pigmentary glaucoma, capsular glaucoma/pseudoexfoliation, or ocular hypertension
* Has been using ocular hypotensive medication on a stable treatment regimen for at least 30 days prior to screening, or is treatment-naive (has never used or has not used ocular hypotensive medication for the last 4 weeks prior to screening)
* Able to discontinue all topical and/or systemic ocular hypotensive medication during the washout period (up to 4 weeks pre-study)
* Best-corrected early treatment of diabetic retinopathy study (ETDRS) visual acuity of 20/80 or better in each eye
* Willing and able to avoid wearing contact lenses from 4 weeks prior to dosing with study medication through 24 hours after final dosing
* Willing and able to self-administer or has an able person available on a daily basis to assist with administration of study medications
* Participant with reproductive potential must agree to remain abstinent (unless abstinence is not a locally acceptable method of contraception) or use highly effective methods of birth control (hormonal contraceptives, intrauterine device, diaphragm, condoms and vasectomy) within the projected duration of the study
* Able to refrigerate study drug at home.

Exclusion Criteria:

* Mean IOP >36 mmHg in either eye at screening
* Unable to use study medication in the affected eye(s)
* History of any inflammatory ocular surface disease or a history of anterior or posterior uveitis in either eye within 6 months prior to screening
* History of retinal detachment, proliferative diabetic retinopathy, or any progressive retinal disease
* Significant visual field loss or evidence of progressive visual loss within the last year
* Intraocular surgery in either eye in the last 4 months
* Any glaucoma surgery, refractive surgery, or penetrating keratoplasty in either eye
* Currently on two or more anti-glaucoma medications (except Cosopt™ or its generic formulation)
* Previously used tafluprost
* History of cardiovascular disorder within 6 months of screening
* History of bronchial asthma, wheezing, chronic obstructive pulmonary disease (COPD) or other pulmonary disease, abnormal chest x-ray, or has current active pneumonia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2013-05-09 (Actual); Study Completion 2013-05-09 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Chabi A, Baranak C, Lupinacci R, Herring WJ. Preservative-free tafluprost in the treatment of open-angle glaucoma or ocular hypertension in India: a phase III clinical trial. Int J Clin Pract. 2016 Jul;70(7):577-86. doi: 10.1111/ijcp.12815. Epub 2016 Jun 13. PMID 27292765
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=2452-002&kw=2452-002&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Tafluprost: One drop of preservative-free vehicle (contains no active drug) per eye in the morning, and one drop of preservative-free tafluprost (0.0015%) per eye in the evening for four weeks.
Period: Overall Study
Arm/Group | Tafluprost | Timolol
Started | 95 | 95
Treated | 93 (The 2 out of 95 started who did not take study drug discontinued due to "Withdrawal by Subject") | 94 (The 1 out of 95 started who did not take study drug discontinued due to "Withdrawal by Subject")
Completed | 87 | 86
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Adverse Event | 3 | 2

BASELINE CHARACTERISTICS:
Population: All Participants as Treated (APaT) population: All randomized participants who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafluprost | Timolol | Total
Number analyzed (Participants) | 93 | 94 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (11.54) | 54.9 (13.42) | 55.8 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 22 | 56
  Male | 59 | 72 | 131
Intraocular Pressure (IOP) - Study Eye [Mean (Standard Deviation); unit: mmHg] — Baseline IOP was measured at 0800, 1000 and 1600 hours; 2 values obtained at each time. If the 2 values differed by ≤2 mmHg, average of 2 was recorded; if by >2 mmHg, a 3rd measurement was made and median of 3 was recorded. Baseline IOP was mean of the values recorded at the 3 time points. One "study eye" was identified, which was the eye with the higher (i.e., "worse") IOP at baseline, or if both eyes had the same baseline IOP value, the right eye was designated the "study eye." Data are for "Per Protocol" population: N=84, 84 and 168 for tafluprost, timolol and Total groups, respectively.
  mmHg | 24.8 (3.0) | 24.9 (2.6) | 24.9 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal IOP Change From Baseline at Week 4 - Study Eye
Description: IOP was measured at baseline, Week 2 and Week 4 using a Goldmann applanation tonometer. At each of these visits, IOP measurement was performed at 0800, 1000 and 1600 hours. At each IOP assessment time point during a visit, 2 consecutive IOP measurements were made. If these 2 measurements differed by ≤2 mmHg, then the average of the 2 IOP values was recorded. If the 2 measurements differed by >2 mmHg, then a third measurement was obtained and the median of these 3 measurements was recorded. The IOP value for a visit (e.g., Week 4) was the mean of the values recorded at the 3 time points during the visit. For each participant, one "study eye" was identified for data summarization and analysis for this primary efficacy outcome measure. The "study eye" was the eye with the higher (i.e., "worse") IOP at baseline, or if both eyes had the same baseline IOP value, the right eye was designated the "study eye." Change from baseline in IOP at Week 4 = Week 4 IOP value - baseline IOP value.
Time Frame: Baseline and Week 4
Population: Per Protocol population: Participants who received at least one dose of study drug, had at least one efficacy measurement available for an analysis endpoint and did not have any protocol violations that may substantially affect the results of the primary efficacy endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Tafluprost | Timolol
Number analyzed (Participants) | 84 | 83
mmHg | -8.3 [-9.0 to -7.6] | -6.6 [-7.3 to -5.9]
Statistical Analysis 1: Comparison: Tafluprost vs Timolol; The study hypothesis was that tafluprost is non-inferior to timolol with respect to change from baseline in diurnal IOP at Week 4 in participants with open-angle glaucoma or ocular hypertension. The study hypothesis would be met if the upper bound of the two-sided 95% confidence interval for the between-treatment difference in mean diurnal IOP change from baseline at Week4 (tafluprost - timolol) was ≤1.5 mmHg; Test type: Non-Inferiority or Equivalence — The study was planned to enroll 248 subjects (124 per treatment group) to yield approximately 230 evaluable subjects (115 per treatment group). The study had power of 90% to test the primary hypothesis. The power and sample size were based on the following assumptions for treatment difference in change from baseline in IOP at Week 4: α = 0.025 (1-sided), Non-inferiority margin = 1.5 mmHg, True treatment difference = 0 mmHg, Standard deviation = 3.5 mmHg; ANCOVA; Analysis model includes terms for treatment, baseline IOP and ocular diagnosis (open-angle glaucoma or ocular hypertension); Difference in Least Squares Means = -1.7, 95% CI 2-sided [-2.6 to -0.7] — Difference is tafluprost - timolol

2. Secondary Outcome: Number of Participants With ≥25% Reduction in IOP From Baseline to Week 4 - Study Eye
Description: IOP was measured at baseline, Week 2 and Week 4 using a Goldmann applanation tonometer. At each of these visits, IOP measurement was performed at 0800, 1000 and 1600 hours. At each IOP assessment time point during a visit, 2 consecutive IOP measurements were made. If these 2 measurements differed by ≤2 mmHg, then the average of the 2 IOP values was recorded. If the 2 measurements differed by >2 mmHg, then a third measurement was obtained and the median of these 3 measurements was recorded. The IOP value for a visit (e.g., Week 4) was the mean of the values recorded at the 3 time points during the visit. For each participant, one "study eye" was identified for data summarization and analysis. The "study eye" was the eye with the higher (i.e., "worse") IOP at baseline, or if both eyes had the same baseline IOP value, the right eye was designated the "study eye." Percent reduction in IOP at Week 4 = ([baseline IOP value - Week 4 IOP value]/Baseline IOP value)*100.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tafluprost | Timolol
Number analyzed (Participants) | 84 | 83
participants | 65 | 48
Statistical Analysis 1: Comparison: Tafluprost vs Timolol; Test type: Superiority or Other; Stratified Miettinen and Nurminen method; Participants were stratified by baseline IOP (<26 mmHg or ≥26 mmHg at 0800 hours) and ocular diagnosis (open-angle glaucoma or ocular hypertension); Difference in percentage = 19.5, 95% CI 2-sided [5.7 to 33.4] — Between-group difference in percentage of participants with ≥25% reduction in IOP at Week 4 = percentage (tafluprost) - percentage (timolol)

3. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Participants with one or more AEs during the study are counted once in this summary.
Time Frame: Up to 14 days after Week 4 visit
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Tafluprost | Timolol
Number analyzed (Participants) | 93 | 94
participants | 28 | 32
Statistical Analysis 1: Comparison: Tafluprost vs Timolol; Test type: Superiority or Other; Miettinen and Nurminen; Difference in percentage = -3.9, 95% CI 2-sided [-17.3 to 9.4] — Between-group difference in percentage of participants with an AE = percentage (tafluprost) - percentage (timolol)

4. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Participants who discontinued study drug treatment due to an AE are counted once in this summary.
Time Frame: Up to Week 4
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Tafluprost | Timolol
Number analyzed (Participants) | 93 | 94
participants | 3 | 2
Statistical Analysis 1: Comparison: Tafluprost vs Timolol; Test type: Superiority or Other; Miettinen and Nurminen; Difference in percentage = 1.1, 95% CI 2-sided [-3.5 to 5.7] — Between-group difference in percentage of participants discontinued study drug due to an AE = percentage (tafluprost) - percentage (timolol)

ADVERSE EVENTS:
Time Frame: Up to 14 days after Week 4 visit
Arm/Group | Tafluprost | Timolol
Serious Adverse Events (participants affected / at risk) | 0/93 | 1/94
Other Adverse Events (participants affected / at risk) | 19/93 | 15/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafluprost (N=93) | Timolol (N=94)
subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafluprost (N=93) | Timolol (N=94)
Conjunctivitis (Eye disorders) | 9 (11) | 9 (10)
Eye irritation (Eye disorders) | 6 (6) | 5 (6)
Eye pruritus (Eye disorders) | 7 (8) | 3 (3)
Ocular hyperaemia (Eye disorders) | 6 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish results for his/her study site after publication of results of entire multicenter trial, or after public disclosure of the results online if a multicenter manuscript is not planned. Sponsor must be able to review all proposed results communications regarding study 60 days prior to submission for publication/presentation. Information identified by the Sponsor as confidential must be deleted prior to submission.